CLINICAL TRIAL: NCT06424782
Title: Investigation of the Therapeutic Effect of the Natural Mineral Water of the Well B-308 OKK in Győr (Gyirmót) Among People With Knee Arthrosis (Randomized, Controlled, Double-blind, Follow-up Study)
Brief Title: Therapeutic Effect of the Natural Mineral Water of the Well B-308 OKK in Győr (Gyirmót) on Knee Osteoarthrosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Collaborators: Gyirmót Sport & Wellness Hotel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-308 OKK
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
Keywords: medicinal water; healing water; balneotherapy; WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicinal water treatment (Experimental): Participants receive medicinal water treatment in bath tub once daily (30 min) on weekdays for 3 weeks.
  Interventions: Other: medicinal water
- Tap water (placebo) treatment (Placebo Comparator): Participants receive placebo water treatment in bath tub once daily (30 min) on weekdays for 3 weeks.
  Interventions: Other: medicinal water

INTERVENTIONS:
Other: medicinal water — Medicinal water treatment in bath tub once daily.

SUMMARY:
The main purpose of the study is to investigate the therapeutic effect of the thermal water of Győr (Gyirmót) well No. B-308 OKK on patients with knee arthrosis, and to compare its therapeutic effect with tap water (placebo) group.

DETAILED DESCRIPTION:
After being informed about the study and the potential risks, all patients giving written informed consent will undergo a continuous screening period, until the number of 25-25 patients is reached, to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 1:1 ratio to medicinal water or placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthrosis that has existed for at least 3 months
* Age between 50 and 80 years
* Willingness to participate in 3-week outpatient rehabilitation treatment
* Pain in the knee joint lasting at least 3 months and at least 5 days a week
* At least mild pain during selection (1 point on the Likert scale)
* Does not have a serious disability

Exclusion Criteria:

* Any kind of physiotherapy treatment in the last 2 months (except home gymnastics)
* Any previous knee joint surgery
* Any trauma to the knee or hip joint in the 1 year prior to the examination
* Knee arthroscopy performed within 3 months prior to the examination
* Intra-articular corticosteroid treatment of the affected knee in the last 3 months
* Palpable Baker's cyst
* Any hip joint or spine surgery within a year before the examination
* Intra-articular hyaluronic injection within 2 months before the examination
* Appearance of lumbar radiculopathy
* Presence of serious internal medicine disease, urogenital or other diseases
* Uncooperative or psychoneurotic patients
* Lumbago, sciatica; and any other surgery or previous fracture in the hip joint
* Subluxation, luxation, algodystrophy, fibromyalgia, gout
* Balneotherapy in the last 6 months
* Systemic corticosteroid treatment in 1 month before the examination
* Starting the treatment of osteoarthritis SYSADOA (symptomatic slow-acting drugs for osteoarthritis) in 3 months before the examination

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in range of motion of the knee measured with goniometer at week 3 and 12 | Baseline and week 3 and 12
  Goniometer is a range of motion measuring device. Its measuring range is 180 degrees. Change = (Week 3 degree - Baseline degree), Change = (Week 12 degree - Baseline degree)
30-second Chair Stand Test | Baseline and week 3 and 12
  The test counts the number of times the patient comes to a full standing position in 30 seconds. Change = (Week 3 number - Baseline number), Change = (Week 12 number - Baseline number)
Timed Up and Go (TUG) | Baseline and week 3 and 12
  It is a simple test that measures how quickly you can stand up, walk 3 meters, turn around, walk back, and sit down. It is done to assess mobility in older adults or predict their risk of falls. Many healthy adults less than 80 years old can complete the TUG test in 10 seconds or less. Change = (Week 3 seconds - Baseline seconds), Change = (Week 12 seconds - Baseline seconds)
Change from baseline in pain on the 10-point Visual Analogue Scale (VAS) at week 3 and 12 | Baseline and week 3 and 12
  The visual analogue scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels. Change = (Week 3 point - Baseline point), Change = (Week 12 point - Baseline point)
Change from baseline in functional status with the Western Ontario and McMaster Universities Arthritis Index (WOMAC) index at week 3 and 12 | Baseline and week 3 and 12
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. The WOMAC is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items). Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status. Change = (Week 3 score - Baseline score), Change = (Week 12 score - Baseline score)
Change from baseline in quality of life with the Short Form 36 Health Survey Questionnaire (SF-36) at week 3 and 12 | Baseline and week 3 and 12
  The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). Scores ranges from 0 to 100. Higher scores indicate higher quality of life. Change = (Week 3 score - Baseline score), Change = (Week 12 score - Baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienn Hanzel, Ph.D., Principal Investigator — University of Pecs
Locations (1):
- Katalin Dr Szendi, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Yes
The outcome measures as individual participant data can be shared. Outcome measures are the followings: range of motion, 30-second Chair Stand Test, Timed Up and Go (TUG), VAS scale, WOMAC index, SF-36 questionnaire
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April 2025 - December 2025
Access Criteria: Data will be provided upon researcher request.

REFERENCES:
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Kulisch A, Benko A, Bergmann A, Gyarmati N, Horvath H, Kranicz A, Mando ZS, Matan A, Nemeth A, Szakal E, Szanto D, Szekeres L, Bender T. Evaluation of the effect of Lake Heviz thermal mineral water in patients with osteoarthritis of the knee: a randomized, controlled, single-blind, follow-up study. Eur J Phys Rehabil Med. 2014 Aug;50(4):373-81. Epub 2014 Mar 5. PMID 24594851
- [Background] Gyarmati N, Kulisch A, Nemeth A, Bergmann A, Horvath J, Mando Z, Matan A, Szakal E, Sasne Peter T, Szanto D, Bender T. Evaluation of the Effect of Heviz Mud in Patients with Hand Osteoarthritis: A Randomized, Controlled, Single-Blind Follow-Up Study. Isr Med Assoc J. 2017 Mar;19(3):177-182. PMID 28457097
- [Background] Ayan C, Carvalho P, Varela S, Cancela JM. Effects of Water-Based Exercise Training on the Cognitive Function and Quality of Life of Healthy Adult Women. J Phys Act Health. 2017 Nov 1;14(11):899-904. doi: 10.1123/jpah.2017-0036. Epub 2017 Sep 25. PMID 28682652
- [Background] Bender T, Balint G, Prohaszka Z, Geher P, Tefner IK. Evidence-based hydro- and balneotherapy in Hungary--a systematic review and meta-analysis. Int J Biometeorol. 2014 Apr;58(3):311-23. doi: 10.1007/s00484-013-0667-6. Epub 2013 May 16. PMID 23677421
- [Background] Karagulle M, Kardes S, Karagulle MZ. Long-term efficacy of spa therapy in patients with rheumatoid arthritis. Rheumatol Int. 2018 Mar;38(3):353-362. doi: 10.1007/s00296-017-3926-8. Epub 2018 Jan 11. PMID 29327104
- [Background] Peter I, Jagicza A, Ajtay Z, Boncz I, Kiss I, Szendi K, Kustan P, Nemeth B. Balneotherapy in Psoriasis Rehabilitation. In Vivo. 2017 Nov-Dec;31(6):1163-1168. doi: 10.21873/invivo.11184. PMID 29102940
- [Background] Gutenbrunner C, Bender T, Cantista P, Karagulle Z. A proposal for a worldwide definition of health resort medicine, balneology, medical hydrology and climatology. Int J Biometeorol. 2010 Sep;54(5):495-507. doi: 10.1007/s00484-010-0321-5. Epub 2010 Jun 9. PMID 20532921
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672